CLINICAL TRIAL: NCT00171366
Title: A Multicenter, Group Study to Evaluate the Safety and Efficacy of Amlodipine and Benazepril Administered in Combination Compared to Amlodipine Monotherapy in Hypertensive Patients Not Adequately Controlled With Amlodipine Alone
Brief Title: A Study Comparing the Response of Patients With Hypertension to Amlodipine or Amlodipine Plus Benazepril.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCIB002H2304
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Hypertension
Keywords: amlodipine; benazepril; hypertension; diastolic
MeSH Terms: conditions — Hypertension; Heart Murmurs | interventions — benazepril

INTERVENTIONS:
Drug: amlodipine/benazepril

SUMMARY:
Comparison of the safety and efficacy of the combination of amlodipine/Benazepril to amlodipine monotherapy in patients with non-essential hypertension, not controlled on amlodipine alone.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 years of age or older.
* Male or female patients are eligible. Female patients must be either post-menopausal for one year or surgically sterile, or using effective, contraceptive methods such as barrier method with spermicide, or an intrauterine device.
* Patients with essential hypertension as measured by a validated device

Exclusion Criteria:

* Severe hypertension (DBP > 115 mmHg diastolic and/or SBP > 180 mmHg systolic).

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1422 (Actual)
Dates: Start 2004-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure at week 6

SECONDARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure at week 6
Change from week 2 in mean sitting diastolic and systolic blood pressure at week 6
Diastolic response rate at week 6. Patients were considered responders if they had a mean sitting diastolic blood pressure of < 90 mmHg or a >= 10 mm Hg decrease compared to baseline.
Change from baseline in 24 hour diastolic and systolic blood pressure at week 6
Change from baseline in 24 hour diastolic and systolic blood pressure at peak which is defined as the lowest hourly blood pressure mean and the average of the hourly means from 4 to 6 hours post dose at week 6

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States